CLINICAL TRIAL: NCT00197678
Title: Comparison of Two Multivitamin Dosage Regimens in the Prevention of Adverse Pregnancy Outcomes Among HIV-Positive Women From Tanzania
Brief Title: Multivitamin Dosage Regimens in the Prevention of Adverse Pregnancy Outcomes Among HIV-Positive Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Wafaie Fawzi MD, DrPH, Harvard School of Public health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HD32257-2
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2010-11

CONDITIONS: HIV Infections
Keywords: HIV; AIDS; Multivitamins; Pregnancy Outcomes; Women; Tanzania; Africa
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multivitamins-Single RDA (Experimental): Multivitamins at doses resembling a single daily Recommended Dietary Allowance (RDA)
  Interventions: Dietary Supplement: Multivitamins-Single RDA
- Multivitamins-Multiples of RDA (Active Comparator): Multivitamin supplements at multiples of the Recommended Dietary Allowance (RDA)
  Interventions: Dietary Supplement: Multivitamins-Multiples of RDA

INTERVENTIONS:
Dietary Supplement: Multivitamins-Multiples of RDA — 20 mg B1, 20 mg B2, 25 mg B6, 50 mcg B12, 100 mg niacin, 500 mg C, 30 mg E, 0.8 mg folic acid taken orally once per day until 6 weeks after delivery
  Arms: Multivitamins-Multiples of RDA
Dietary Supplement: Multivitamins-Single RDA — 1.4 mg B1, 1.4 mg B2, 1.9 mg B6, 50 mcg B12, 100 mg niacin, 70 mg C, 10 mg E, and 0.4 mg folic acid taken orally once per day until 6 weeks after delivery
  Arms: Multivitamins-Single RDA

SUMMARY:
The purpose of this study is to examine effects of daily administration of multivitamin supplements at doses resembling the Recommended Dietary Allowance (RDA) during pregnancy to HIV positive women decreases the risks of low birth weight (<2500 g), and pre-term birth (< 37 weeks gestation), compared to multivitamin supplements at doses above the RDA.

DETAILED DESCRIPTION:
This is a randomized clinical trial conducted to examine effects of daily administration of multivitamin supplements at doses resembling the Recommended Dietary Allowance (RDA) during pregnancy to HIV positive women decreases the risks of low birth weight (<2500 g), and pre-term birth (< 37 weeks gestation), compared to multivitamin supplements at doses above the RDA. All women receive standard prenatal care, including nevirapine for the prevention of mother-to-child transmission of HIV.

ELIGIBILITY:
Inclusion Criteria:

- HIV-positive pregnant women who are between 12 and 27 weeks gestation who intend to stay in Dar es Salaam until delivery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1141 (Actual)
Dates: Start 2002-11; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Low birthweight (< 2500 g) | Delivery
Pre-term birth (< 36 weeks gestation) | Monthly until the 32nd week of pregnancy, once every 2 weeks from 32nd to 36th week

CONTACTS AND LOCATIONS:
Overall Officials: Wafaie W. Fawzi, MD,DrPH, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Harvard School of Public Health, Boston, Massachusetts, United States

REFERENCES:
- [Result] Kawai K, Kupka R, Mugusi F, Aboud S, Okuma J, Villamor E, Spiegelman D, Fawzi WW. A randomized trial to determine the optimal dosage of multivitamin supplements to reduce adverse pregnancy outcomes among HIV-infected women in Tanzania. Am J Clin Nutr. 2010 Feb;91(2):391-7. doi: 10.3945/ajcn.2009.28483. Epub 2009 Nov 25. PMID 19939985